CLINICAL TRIAL: NCT03507153
Title: Muscle Activity Evaluation of Maxillary Bilateral Bounded Partial Denture Fabricated By Bre-Flex Versus Peek (Randomized Clinical Trial)
Brief Title: Muscle Activity Evaluation of Maxillary Bilateral Bounded Partial Denture Fabricated By Bre-Flex Versus Peek
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed salama sayed tantawy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ASalama
Record Dates: First submitted 2018-03-23; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Maxillary Class III Modification I Edentulous Patients
Keywords: "Nylon denture base" and "PEEK partial denture"

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Only statistician will be blinded as the 2 materials have different colors The patients: they won't be aware of the lab procedures till finishing and delivery of the dentures.
  The outcome assessor: the assessor who will assess the muscular activity will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bre-fllex group (Active Comparator): Maxillary class III modification I edentulous patients that will recieve Bre-flex partial denture
  Interventions: Procedure: Bre-flex maxillary partial denture
- PEEK group (Experimental): Maxillary class III modification I edentulous patients that will recieve PEEK partial denture
  Interventions: Procedure: PEEK maxillary partial denture

INTERVENTIONS:
Procedure: Bre-flex maxillary partial denture — Partial denture fabricated from Bre.flex material.
  Arms: Bre-fllex group
Procedure: PEEK maxillary partial denture — Partial denture fabricated from PEEK material.
  Arms: PEEK group

SUMMARY:
Evaluation of the muscle activity of masseter in tooth borne partial denture wearers (class III modification 1 Kennedy's classification) with two different denture base materials (Breflex and PEEK) by means of electromyograph.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have Kennedy class III modification I upper partially edentulous ridges.
* The remaining teeth have good periodontal condition, with no signs of attrition or gingival recession.
* All patients have skeletal Angle's class I maxillo-mandibular relationship and have sufficient interarch distance.
* Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.
* Free from any tempro-mandibular joint disorder.
* The patients have good oral hygiene and low caries index.

Exclusion Criteria:

* Patients having abnormal habits as bruxism or clenching.
* Patients having hormonal disorders as diabetes, thyroid or parathyroid hormonal diseases were not included.
* Teeth with compromised bone support.
* Patient with xerostomia or excessive salivation.
* Patient with abnormal tongue behavior and/or size.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Muscular activity | one month
  Evaluation of the muscle activity of masseter in tooth borne partial denture wearers (class III modification 1 Kennedy's classification) with two different denture base materials (Breflex and PEEK) by means of electromyograph.

IPD SHARING:
Plan to Share IPD: No